CLINICAL TRIAL: NCT05650879
Title: A Phase 1a/1b Study of ELVN-002 for the Treatment of Patients With HER2 Mutant Non-Small Cell Lung Cancer
Brief Title: ELVN-002 in HER2 Mutant Non-Small Cell Lung Cancer
Acronym: HER2
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Enliven Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ELVN-002-001
Record Dates: First submitted 2022-11-28; First posted 2022-12-14 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: HER2 Mutant Non-small Cell Lung Cancer; HER2-positive Metastatic Breast Cancer; HER2 Gene Mutation; HER2 Amplification
Keywords: HER2 genetic alterations; HER2 mutation; ELVN-002; Non-small cell lung cancer; HER-2 positive metastatic breast cancer; Enhertu; trastuzumab emtansine; fam-trastuzumab deruxtecan-nxki; Kadcyla
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Ado-Trastuzumab Emtansine

STUDY DESIGN:
Intervention Model Description: Phase 1 will be a dose escalation monotherapy according to the Bayesian Optimal Interval Design model Phase 1b will be a dose expansion: up to 40 patients randomized between 2 dose levels
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Phase 1a Monotherapy Dose Escalation (Experimental): ELVN-002 will be administered either once or twice daily. Each cohort of patients will receive a higher dose. ELVN-002 is an oral capsule. Duration of treatment will be until disease progression or patient discontinues ELVN-002 for another reason.
  Interventions: Drug: ELVN-002
- Phase 1a Monotherapy Dose Exploration (Experimental): ELVN-002 will be administered either once or twice daily. A maximum of 80 patients will enroll in this arm. A maximum of 10 patients may be enrolled at a single dose or tumor type. ELVN-002 is an oral capsule. Duration of treatment will be until disease progression or patient discontinues ELVN-002 for another reason.
  Interventions: Drug: ELVN-002
- Phase 1b Monotherapy Dose Expansion (Experimental): ELVN-002 will be administered either once or twice daily. A maximum of 40 patients will enroll in this arm. Patients will be randomized 1:1 to one of two dose levels.
  ELVN-002 is an oral capsule. Duration of treatment will be until disease progression or patient discontinues ELVN-002 for another reason.
  Interventions: Drug: ELVN-002
- Phase 1a Combination Dose Escalation with T-DXd (Experimental): ELVN-002 will be administered either once or twice daily starting on Day 1. ELVN-002 is an oral capsule. Each cohort will receive a higher dose of ELVN-002. All patients in all cohorts will initiate with 5.4mg/kg of intravenous T-DXd once every 3 weeks starting on day 22 of the study. Duration of treatment will be until disease progression or patient discontinues ELVN-002 for another reason.
  Interventions: Drug: ELVN-002; Drug: Fam-Trastuzumab Deruxtecan-Nxki
- Phase 1a Combination Dose Escalation with T-DM1 (Experimental): ELVN-002 will be administered either once or twice daily starting on Day 1. ELVN-002 is an oral capsule. Each cohort will receive a higher dose of ELVN-002. All patients in all cohorts will initiate with 3.6 mg/kg of intravenous T-DM1 once every 3 weeks starting on day 22 of the study. Duration of treatment will be until disease progression or patient discontinues ELVN-002 for another reason.
  Interventions: Drug: ELVN-002; Drug: Trastuzumab emtansine

INTERVENTIONS:
Drug: ELVN-002 — capsule
Drug: Fam-Trastuzumab Deruxtecan-Nxki — intravenous
  Other Names: Enhertu; T-DXd
  Arms: Phase 1a Combination Dose Escalation with T-DXd
Drug: Trastuzumab emtansine — intravenous
  Other Names: Kadcyla; T-DM1
  Arms: Phase 1a Combination Dose Escalation with T-DM1

SUMMARY:
The goal of this clinical trial is to test ELVN-002 in people with cancers that have an abnormal HER2 gene. The main question the trial aims to answer is if ELVN-002 is safe and tolerable at different doses. A second main question is to evaluate the concentration of ELVN-002 in the blood at different doses and to see how this correlates with safety and see how the concentration of drug changes over time. The third main question is to see if ELVN-002 works to shrink cancers that have HER2 genetic abnormalities, particularly non-small cell lung cancer.

DETAILED DESCRIPTION:
There are 4 parts to the trial. Part 1 is a dose escalation with ELVN-002 monotherapy for people with advanced stage solid tumors that have a HER2 mutation, amplification or high HER2 over-expression. Part 2 is an ELVN-002 monotherapy dose exploration where additional people may be enrolled at dose levels that have cleared the dose escalation in Part 1 to further evaluate the safety, tolerability, pharmacokinetics and clinical activity. Part 3 is a dose expansion of ELVN-002 monotherapy which will enroll up to 40 patients people with advanced stage HER2 mutant non-small cell lung cancer. Patients in Part 3 will be randomized 1:1 to receive one of two dose levels.

Part 4 is a combination dose escalation where, based on the results of Part 1 and 2, a combination of ELVN-002 and either fam-trastuzumab deruxtecan-nxki (in HER2 mutant non-small cell lung cancer) or trastuzumab emtansine (in HER2 positive breast cancer) will be evaluated for safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

Phase 1a Monotherapy Dose Escalation and Exploration:

* Pathologically documented advanced stage solid tumor
* Progressed following all standard treatment or not appropriate for standard treatment
* HER2 mutation, HER2 amplification or HER2 positive based on local testing

Phase 1b Monotherapy

* Pathologically documented unresectable and/or metastatic non-squamous NSCLC
* HER2 mutation identified by tissue (fresh or archival) or ctDNA. Local testing for up to 20 patients the remainder centrally confirmed.
* Measurable disease
* No known epidermal growth factor receptor (EGFR), ROS1, anaplastic lymphoma kinase (ALK), or BRAF V600E mutation
* Progressed after receiving at least 1 prior systemic therapy including a platinum-based chemotherapy with or without immunotherapy, or not appropriate for standard treatment.
* No prior HER2 tyrosine kinase inhibitor. Prior HER2 directed antibodies or anti-body drug conjugates are allowed
* No limit on prior number of therapies

Phase 1a Combination with T-DXd

* Pathologically documented advanced stage NSCLC
* Progressed after receiving at least 1 prior systemic therapy.
* HER2 mutation based on local/historical testing of tissue or circulating tumor DNA
* No known EGFR, ROS1, ALK, or BRAF V600E mutation
* No prior T-DXd
* No clinically severe pulmonary compromise
* No limit on prior number of therapies

Phase 1a Combination Breast Cancer

* Documented HER2 positive (Immunohistochemical [IHC] 3+ or IHC2+/in situ hybridization (ISH+) breast cancer
* Must have previously received trastuzumab, a taxane, and T-DXd (if available and appropriate) in the metastatic setting.
* No limit on prior number of therapies
* No prior T-DM1

All Phases

* Eastern Cooperative Oncology Group performance status of 0-1
* Left ventricular ejection fraction ≥ 50%
* Platelet count ≥ 100 x 109/L
* Hemoglobin ≥ 8.5 g/dL
* Absolute neutrophil count ≥1.0 x 109/L
* Total bilirubin < 1.5 times upper limit of normal range (ULN), except for patients with Gilbert's syndrome
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) < 3 times ULN. In the setting of liver metastases < 5 times ULN.
* Creatinine clearance ≥ 60 mL/minute

Exclusion Criteria All Phases:

* Severe cardiac arrhythmias, requiring treatment, symptomatic congestive heart failure, myocardial infarction within 28 days prior to first dose, or unstable angina.
* Another active malignancy within 2 years except basal cell skin cancer and carcinoma in situ treated curatively
* Active or chronic liver disease
* Active infection requiring systemic therapy within 14 days before the first dose
* Brain lesion requiring immediate local therapy
* Leptomeningeal disease
* Uncontrolled seizures
* Corrected QT interval (QTc) of >470 milliseconds (ms) females or >450 ms for males by Fridericia (QTcF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities in Phase 1a monotherapy | 21 days
Incidence of adverse events in Phase 1a monotherapy | 24 months
incidence of laboratory abnormalities in Phase 1a monotherapy | 24 months
incidence of ECG abnormalities in Phase 1a monotherapy | 24 months
incidence of dose limiting toxicities in Phase 1a combination with fam-trastuzumab deruxtecan (T-DXd) | 42 days
Incidence of adverse events in Phase 1a combination with T-DXd | 24 months
incidence of laboratory abnormalities in Phase 1a combination with T-DXd | 24 months
incidence of ECG abnormalities in Phase 1a combination with T-DXd | 24 months
incidence of dose limiting toxicities in Phase 1a combination with trastuzumab emantasine (T-DM1) | 42 days
Incidence of adverse events in Phase 1a combination with T-DM1 | 24 months
incidence of laboratory abnormalities in Phase 1a combination with T-DM1 | 24 months
incidence of ECG abnormalities in Phase 1a combination with T-DM1 | 24 months
Incidence of adverse events in Phase 1b monotherapy | 24 months
incidence of laboratory abnormalities in Phase 1b monotherapy | 24 months
incidence of ECG abnormalities in Phase 1b monotherapy | 24 months

SECONDARY OUTCOMES:
Objective Response rate in Phase 1a monotherapy | 24 months
  For patients with measurable disease at baseline, confirmed response per RECIST 1.1
Objective response rate in Phase 1b monotherapy | 24 months
  Confirmed response per RECIST 1.1
Duration of response in Phase 1b monotherapy | 24 months
  The time from the first response to progression or death per RECIST 1.1
Brain metastases response in Phase 1b monotherapy | 24 months
  for patients with measurable brain metastases at baseline, the percent of patients who have a confirmed response per RECIST 1.1
PK parameter of area under the curve of ELVN-002 in Phase 1a monotherapy | 21 days
  the concentration of ELVN-002 measured in the blood over 24 hours at steady state
PK parameter of maximum concentration of ELVN-002 in Phase 1a monotherapy | 21 days
  the maximum concentration of ELVN-002 measured in the blood at any time point at steady state
PK parameter of terminal half life of ELVN-002 in Phase 1a monotherapy | 21 days
  the half life of ELVN-002 calculated from the concentration of ELVN-002 in blood
PK parameter of area under the curve of ELVN-002 in Phase 1b monotherapy | 21 days
  the concentration of ELVN-002 measured in the blood over 24 hours at steady state
PK parameter of maximum concentration of ELVN-002 in Phase 1b monotherapy | 21 days
  the maximum concentration of ELVN-002 measured in the blood at any time point at steady state
PK parameter of terminal half life of ELVN-002 in Phase 1b monotherapy | 21 days
  the half life of ELVN-002 calculated from the concentration of ELVN-002 in blood

CONTACTS AND LOCATIONS:
Locations (39):
- United States (5):
  - University of Colorado - Anschutz Medical Campus - PPDS, Aurora, Colorado
  - Advent Health Orlando, Orlando, Florida
  - BRCR Medical Center Inc, Plantation, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - NEXT/Virginia Cancer Specialists, Fairfax, Virginia
- Australia (3):
  - Macquarie University Hospital, Westmead, New South Wales
  - Linear Clinical Research Limited, Nedlands, Western Australia
  - Blacktown Hospital, Darlinghurst
- France (7):
  - Hôpital de la Timone Centre d'essais en cancérologie de Marseille (CEPCM-CLIPP), Marseille, Bouches-du-Rhône
  - Hôpital Pontchaillou, Rennes, Brittany Region
  - Centre Francois Baclesse, Caen, Calvados
  - EDOG - Institut Bergonie - PPDS, Bordeaux, Gironde
  - Centre Georges François Leclerc, Dijon
  - Centre Léon Berard, Lyon
  - Institut Gustave Roussy (IGR), Villejuif
- Italy (6):
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Lombardy
  - Fondazione del Piemonte per l'Oncologia (IRCCS), Candiolo, Piedmont
  - SOC Oncologia Medica e dei Tumori lmmunocorrelati, Centro Di Riferimento Oncologico Di Aviano (CRO) IRCCS, Aviano, Pordenone
  - Azienda Ospedaliero Universitaria delle Marche, Ancona, The Marches
  - Fondazione Policlinico Universitario A. Gemelli, Roma
  - Unità Operativa Oncologia medica ed Ematologia, Rozzano
- South Korea (6):
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggido
  - Gachon University Gil Medical Center, Incheon
  - Severence Hospital, Yonsei University, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
- Spain (9):
  - Hospital Universitari Arnau de Vilanova, Lleida, Lleida
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - START Barcelona Hospital HM Nou Delfos, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - lnstitut Catala d'Oncologia (ICO) L'Hospitalet, Servicio de Oncologia Medica, L'Hospitalet de Llobregat
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Fundación Instituto Valenciano de Oncología, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia
- Taiwan (3):
  - Taichung Veterans General Hospital, Taichung
  - National Chen Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No